CLINICAL TRIAL: NCT03068949
Title: A Comparison of CD4 T Cell Induction and Antibody Responses Between a Pure Hemagglutinin Influenza Vaccine and Licensed Subvirion Influenza Vaccine Made in Eggs or Cell Culture in Healthy Adults.
Brief Title: Comparison of Three Licensed Influenza Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Angela Branche, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 59331; 272201400005C-P00019-9999-4 (NIH)
Record Dates: First submitted 2017-02-23; First posted 2017-03-03 (Actual); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluBlok; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- FluBlok (Active Comparator): FluBlok 0.5 mL given IM X1
  Interventions: Biological: FluBlok
- Fluzone (Active Comparator): Fluzone 0.5 mL given IM X1
  Interventions: Biological: Fluzone
- FluCelVax (Active Comparator): FluCelVax 0.5 mL given IM X 1
  Interventions: Biological: FluCelVax
- Fluzone HD (Active Comparator): Fluzone HD 0.5 mL given IM X1
  Interventions: Biological: Fluzone HD

INTERVENTIONS:
Biological: FluBlok — FluBlok trivalent Influenza Vaccine .5 mL given Intramuscularly
  Arms: FluBlok
Biological: Fluzone — Fluzone Quadrivalent Influenza Vaccine .5 mL given intramuscularly
  Arms: Fluzone
Biological: FluCelVax — FluCelVax Quadrivalent Influenza Vaccine .5 mL given intramuscularly
  Arms: FluCelVax
Biological: Fluzone HD — Fluzone HD Trivalent High Dose Influenza Vaccine .5 mL given intramuscularly
  Arms: Fluzone HD

SUMMARY:
This study will evaluate in detail the way that the immune system responds to three different kinds of flu shots that are licensed in the United States.

DETAILED DESCRIPTION:
Previous observations to date lead to the following model: Traditional egg-derived TIV have contaminating internal virion proteins that preferentially elicit memory CD4 T cells specific for these proteins. These CD4 T cells will have limited efficacy as helpers for the neutralizing Ab response and will suppress the CD4 T cell response to new HA epitopes in the vaccine. The current study will test this hypothesis by comparing CD4 cell responses to specific epitopes, and the subsequent B cell and antibody response, in subjects receiving a vaccine containing only HA protein to vaccines with more complex antigenic characteristics. The CD4 T cell reactivity to pools of unique, conserved, and total pH1 HA peptides as well as H3, influenza B HA, NP, and M1 peptides will be quantified using cytokine Elispot assays and flow cytometry, and then compared to the subsequent antibody and B cell response.

Investigators will also use this study as an opportunity to evaluate the effects of prior vaccination. Recent studies have emphasized the potential negative effect of vaccination in prior years on both the immune response as well as the protective effectiveness of current vaccine. In order to evaluate this phenomenon in the context of multiple vaccine formulations, prior vaccination history of the subjects will be reviewed and subjects stratify vaccination based on vaccine history.

In addition, subjects who participated in this study in a previous year are eligible to re-enroll, and will receive the same vaccine that they were randomized to previously. This will allow an evaluation of differences between vaccine formulations in the responsiveness to multiple vaccinations.

Furthermore, recent studies indicate reports that the glycosylation pattern of viral hemagglutinins produced in cell culture can vary depending on the host cell used, and that this can affect CD4 T cell immunogenicity and antibody recognition. As a cell culture-based influenza vaccine production platform offers many advantages and may eventually supplant the traditional egg-based approach, it is of great value to understand the CD4 T cell response induced by this vaccine and how this affects neutralizing Ab production.

Recent data have also suggested that the failure of seasonal influenza infection to induce substantial levels of stalk specific antibody may be due to the relatively inaccessible nature of this epitope. As part of this study, investigators will also compare the specificity of the human antibody response between the vaccine groups, with the hypothesis that the rHA vaccine will more readily allow targeting of these important, broadly conserved epitopes. There is compelling preliminary data demonstrating that multiple antibodies that we have isolated have a particularly slow on rate when they bind to the HA-stalk versus the HA-globular head epitopes on whole virions, but not on recombinant HA trimmers expressed in baculovirus. The hypothesis is that a free, recombinant HA vaccine will allow more efficient targeting of the HA-Stalk epitopes.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 49 years of age (inclusive).
2. Female subjects must fulfill one of the following: (i) not able to bear children because she has been surgically sterilized (tubal ligation or hysterectomy) or (ii) agrees to practice effective methods of contraception that may include, but are not limited to abstinence, barrier methods, monogamous relationship with vasectomized partner, birth control pills, patches, hormonal shots or hormonal implants, NuvaRing and IUDs (intrauterine devices), from 30 days prior to study enrollment through 30 days following receipt of the last dose of vaccine.
3. Female subjects of childbearing potential must have a negative pregnancy test (urine or serum) within 24 hours prior to vaccination.
4. The subject must be in good health, as determined by: vital signs (heart rate >55 to <100 bpm; blood pressure: systolic ≥ 90 mm Hg and ≤150 mm Hg; diastolic ≤ 90 mm Hg; oral temperature <100.0ºF); medical history; and targeted physical examination, when necessary, based on medical history. Stable medical condition is defined as: no recent increase in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months.
5. The subject is able to understand and comply with the planned study procedures, including being available for all study visits.
6. The subject has provided informed consent prior to any study procedures.
7. Subjects who have not received seasonal flu vaccine for the current year.

Exclusion Criteria

1. Subject report of known hypersensitivity to allergy to components of the study vaccine or other components of the study vaccine.
2. Subject report of known latex allergy
3. Subject report of a history of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines.
4. Subject report of a history of Guillain-Barre syndrome within 6 weeks of receipt of a previous influenza vaccine.
5. The subject is a woman who is pregnant or breastfeeding or intends to become pregnant during the study period between enrollment and 30 days following receipt of vaccine.
6. The subject is immunosuppressed as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
7. The subject has an active neoplastic disease (excluding non-melanoma skin cancer or prostate cancer that is stable in the absence of therapy) or a history of any hematological malignancy. For this criterion, "active" is defined as having received treatment within the past 5 years.
8. The subject has long-term (greater than 2 weeks) use of oral or parenteral steroids, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (nasal and topical steroids are allowed).
9. The subject received immunoglobulin or another blood product within the 3 months prior to enrollment in this study.
10. The subject has received an inactivated vaccine within the 2 weeks or a live vaccine within the 4 weeks prior to enrollment in this study or plans to receive another vaccine within the next 28 days.
11. The subject has an acute or chronic medical condition that, in the opinion of the investigator or appropriate sub-investigator, would render vaccination unsafe or would interfere with the evaluation of responses. These conditions include any acute or chronic medical disease or conditions defined as persisting for 3 months (defines ad 90 days) or longer, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses of the subject's successful completion of the study.
12. Subjects with an active infection or that has an acute illness or an oral temperature greater than 99.9F (37.7C) within 3 days prior to enrollment or vaccination. Subjects who had an acute illness that was treated symptoms resolved are eligible to enroll as long as treatment is completed and symptoms resolved > 3 days prior to enrollment.
13. The subject is currently participating or plans to participate in a study that involves an experimental agent (vaccine, drug, biologic, device, blood product, or medication) or has received an experimental agent within 1 month prior to enrollment in this study, or expects to receive another experimental agent during participation in this study, or intends to donate blood during the study period.
14. The subject has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
15. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
16. The subject has a diagnosis of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis, or is receiving psychiatric drugs. Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment without decompensation are allowed enrollment into the study.
17. The subject has a history of alcohol or drug abuse in the 5 years prior to enrollment.
18. The subject has a known human immunodeficiency virus, hepatitis B, or hepatitis C infection.
19. The subject has any condition that the principal investigator (PI) believes may interfere with successful completion of the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 413 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Branche, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Vaccine Research Unit Room 3-5000, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the CEIRS (Centers of Excellence for Influenza Research and Surveillance) network
Supporting Information: Study Protocol
Time Frame: 12 months
Access Criteria: Broad Access

REFERENCES:
- [Derived] Gouma S, Zost SJ, Parkhouse K, Branche A, Topham DJ, Cobey S, Hensley SE. Comparison of Human H3N2 Antibody Responses Elicited by Egg-Based, Cell-Based, and Recombinant Protein-Based Influenza Vaccines During the 2017-2018 Season. Clin Infect Dis. 2020 Sep 12;71(6):1447-1453. doi: 10.1093/cid/ciz996. PMID 31598646

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FluBlok | Fluzone | FluCelVax | Fluzone HD
Started | 113 | 102 | 122 | 76
Completed | 105 | 90 | 113 | 63
Not Completed | 8 | 12 | 9 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FluBlok | Fluzone | FluCelVax | Fluzone HD | Total
Number analyzed (Participants) | 113 | 102 | 122 | 76 | 413
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (16.7) | 29.0 (10.2) | 33.4 (15.6) | 35.9 (18.0) | 33.0 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 52 | 67 | 39 | 230
  Male | 41 | 50 | 55 | 37 | 183
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 11 | 5 | 22
  Not Hispanic or Latino | 112 | 97 | 111 | 71 | 391
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change of HAI Serum Antibody Titers to A/California/07/09 (H1N1)
Description: Mean change of HAI serum antibody titers to A/California/07/09 (H1N1) using serum hemagglutination-inhibition (HAI) assay.
Time Frame: Day 0 to Day 28
Population: HAI serum antibody titers to A/California/07/09 (H1N1) for Fluzone HD arm are unavailable. Fluzone HD group was only enrolled in flu seasons Fall 2017 - Fall 2019. HAI serum antibody titers to A/California/07/09 (H1N1) was only tested on subjects enrolled in Fall 2015 and Fall 2016.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | FluBlok | Fluzone | FluCelVax
Number analyzed (Participants) | 32 | 31 | 38
titer | 1937 [636 to 3238] | 383 [176 to 590] | 607 [370 to 845]

2. Primary Outcome: Mean Change of HAI Serum Antibody Titers to A/Michigan/45/2015 (H1N1)
Description: Mean Change of HAI Serum Antibody Titers to A/Michigan/45/2015 (H1N1) using serum hemagglutination-inhibition (HAI) assay.
Time Frame: Day 0 to Day 28
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | FluBlok | Fluzone | FluCelVax | Fluzone HD
Number analyzed (Participants) | 23 | 25 | 30 | 22
titer | 564 [68 to 1059] | 420 [137 to 703] | 354 [143 to 564] | 898 [238 to 1557]

3. Primary Outcome: Mean Change of HAI Serum Antibody Titers to A/Switzerland/9715293/13 (H3N2)
Description: Mean Change of HAI Serum Antibody Titers to A/Switzerland/9715293/13 (H3N2)
Time Frame: Day 0 to Day 28
Population: HAI serum antibody titers to A/Switzerland/9715293/13 (H3N2) for Fluzone HD arm are unavailable. Fluzone HD group was only enrolled in flu seasons Fall 2017 - Fall 2019. HAI serum antibody titers to A/Switzerland/9715293/13 (H3N2) was only tested on subjects enrolled in Fall 2015 and Fall 2016.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | FluBlok | Fluzone | FluCelVax
Number analyzed (Participants) | 32 | 31 | 38
titer | 1733 [655 to 2811] | 1711 [450 to 2971] | 799 [221 to 1377]

4. Primary Outcome: Mean Change of MN Serum Antibody Titers to A/California/07/09 (H1N1)
Description: Mean Change of MN Serum Antibody Titers to A/California/07/09 (H1N1) using Microneutralization (MN) assay.
Time Frame: Day 0 to Day 28
Population: MN serum antibody titers to A/California/07/09 (H1N1) for Fluzone HD arm are unavailable. Fluzone HD group was only enrolled in flu seasons Fall 2017 - Fall 2019. MN serum antibody titers to A/California/07/09 (H1N1) was only tested on subjects enrolled in Fall 2015 and Fall 2016.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | FluBlok | Fluzone | FluCelVax
Number analyzed (Participants) | 32 | 31 | 38
titer | 2786 [1390 to 4182] | 373 [131 to 615] | 881 [477 to 1286]

5. Primary Outcome: Mean Change of MN Serum Antibody Titers to A/Michigan/45/2015 (H1N1)
Description: Mean Change of MN Serum Antibody Titers to A/Michigan/45/2015 (H1N1) using Microneutralization (MN) assay.
Time Frame: Day 0 to Day 28
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | FluBlok | Fluzone | FluCelVax | Fluzone HD
Number analyzed (Participants) | 23 | 25 | 30 | 22
titer | 1007 [246 to 1769] | 554 [104 to 1003] | 308 [94 to 710] | 1477 [660 to 2293]

6. Primary Outcome: Mean Change in CD4 T Cells Reactivity to Pools of Total pHA Peptides Derived From pH1N1 HA
Description: Mean change in CD4 T cells reactivity to pools of total pHA peptides derived from pH1N1 HA using cytokine Elispot
Time Frame: Day 0 to Day 14
Measure: Mean (Standard Error); unit: cells per million CD8- and CD56- PBMC
Arm/Group | FluBlok | Fluzone | FluCelVax | Fluzone HD
Number analyzed (Participants) | 50 | 49 | 51 | 21
cells per million CD8- and CD56- PBMC | 71.2 (97.4) | 21.4 (57.3) | 29.5 (92.8) | 39.8 (84.7)

7. Primary Outcome: Mean Change in CD4 T Cells Reactivity to Pools of Total pHA Peptides Derived From H3 HA
Description: Mean change in CD4 T cells reactivity to pools of total pHA peptides derived from H3 HA using cytokine Elispot
Time Frame: Day 0 to Day 14
Measure: Mean (Standard Error); unit: cells per million CD8- and CD56- PBMC
Arm/Group | FluBlok | Fluzone | FluCelVax | Fluzone HD
Number analyzed (Participants) | 50 | 49 | 51 | 21
cells per million CD8- and CD56- PBMC | 93.2 (128.0) | 14.0 (69.8) | 21.5 (157.3) | 58.6 (162.7)

8. Primary Outcome: Mean Change in CD4 T Cells Reactivity to Pools of Total pHA Peptides Derived From Influenza B HA
Description: Mean change in CD4 T cells reactivity to pools of total pHA peptides derived from influenza B HA using cytokine Elispot.
Time Frame: Day 0 to Day 14
Measure: Mean (Standard Error); unit: cells per million CD8- and CD56- PBMC
Arm/Group | FluBlok | Fluzone | FluCelVax | Fluzone HD
Number analyzed (Participants) | 50 | 49 | 51 | 21
cells per million CD8- and CD56- PBMC | 178.0 (218.8) | 89.2 (162.1) | 79.0 (203.5) | 42.1 (171.6)

9. Primary Outcome: Mean Change in CD4 T Cells Reactivity to Pools of Total pHA Peptides Derived From NP
Description: Mean change in CD4 T cells reactivity to pools of total pHA peptides derived from NP using cytokine Elispot.
Time Frame: Day 0 to Day 14
Measure: Mean (Standard Error); unit: cells per million CD8- and CD56- PBMC
Arm/Group | FluBlok | Fluzone | FluCelVax | Fluzone HD
Number analyzed (Participants) | 49 | 49 | 51 | 20
cells per million CD8- and CD56- PBMC | -23.9 (81.3) | -9.7 (95.5) | -16.9 (128.1) | 19.6 (165.2)

10. Primary Outcome: Mean Change in CD4 T Cells Reactivity to Pools of Total pHA Peptides Derived From M1
Description: Mean change in CD4 T cells reactivity to pools of total pHA peptides derived from M1 using cytokine Elispot.
Time Frame: Day 0 to Day 14
Measure: Mean (Standard Error); unit: cells per million CD8- and CD56- PBMC
Arm/Group | FluBlok | Fluzone | FluCelVax | Fluzone HD
Number analyzed (Participants) | 50 | 49 | 51 | 21
cells per million CD8- and CD56- PBMC | -18.9 (99.7) | -18.7 (118.0) | 20.9 (143.8) | -36.3 (212.3)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | FluBlok | Fluzone | FluCelVax | Fluzone HD
All-Cause Mortality (participants affected / at risk) | 0/113 | 0/102 | 0/122 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/113 | 0/102 | 0/122 | 0/76
Other Adverse Events (participants affected / at risk) | 36/113 | 30/102 | 45/122 | 28/76
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FluBlok (N=113) | Fluzone (N=102) | FluCelVax (N=122) | Fluzone HD (N=76)
abdomina l pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
bilateral conjunctivities (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
body aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
chipped tooth/dentral extraction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
concussion (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (4) | 0 (0)
Uri (Respiratory, thoracic and mediastinal disorders) | 18 (21) | 21 (21) | 24 (26) | 14 (17)
sore throat (General disorders) | 1 (1) | 3 (3) | 4 (4) | 3 (3)
sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
strep throat (Infections and infestations) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
urinary tract infection (Infections and infestations) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
yeast infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
tooth ache (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
serous otitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
influenza like illness (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
influenza (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
feverish (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
headache (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
myalgia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
injection site bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
injection site erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
injection site hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
injection site pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
injection site swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
foot pain due to bone chip (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
fractured right thumb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
knee replacement surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
left wrist pain secondary to electric shock (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
left arm pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
left arm laceration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
right ankle sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
right elbow pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
sensation of heaviness and heat of legs (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
tendon sheath inflammation (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dizziness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
trembling in hands (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
migraine headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
tingling in both hands (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
lethargy (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
lightheadedness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
sneezing (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
rhinitis (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
gastrointestional illness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
stomach ache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
rigth breast lump (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
right ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
eyelid swelling (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
heart palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
thyroid nodules (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
vaginal spotting (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
right labral pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/49/NCT03068949/Prot_SAP_000.pdf